CLINICAL TRIAL: NCT04064047
Title: Anorectal Application of 5% Lidocaine Cream Reduces Pain Prior to Periprostatic Nerve Block During Transrectal Ultrasound Guided Biopsy: Randomized, Prospective Controlled Study
Brief Title: Anorectal Application of 5% Lidocaine Cream Reduces Pain Prior to Periprostatic Nerve Block During Transrectal Ultrasound Guided Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: Assaf-HarofehMC 0289-15-ASF
Record Dates: First submitted 2019-01-20; First posted 2019-08-21 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Pain; Prostate Cancer; Rectal/Anal
MeSH Terms: conditions — Pain; Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- External Anal application - 5 minutes exposure (Active Comparator): Anal application of lidocaine cream 5% for 5 minutes before probe insertion. After probe insertion and prior to biopsy, a periprostatic nerve block was performed with 10 mL of 1% Lidocaine (5 mL on each side).
  Interventions: Procedure: Trans rectal ultrasound guided prostate biopsy; Procedure: Trans rectal ultrasound; Procedure: Prostate biopsy; Procedure: Periprostatic nerve block
- External Anal application - 10 minutes exposure (Active Comparator): Anal application of lidocaine cream 5% for 10 minutes before probe insertion. After probe insertion and prior to biopsy, a periprostatic nerve block was performed with 10 mL of 1% Lidocaine (5 mL on each side).
  Interventions: Procedure: Trans rectal ultrasound guided prostate biopsy; Procedure: Trans rectal ultrasound; Procedure: Prostate biopsy; Procedure: Periprostatic nerve block
- External Anal application - 20 minutes exposure (Active Comparator): Anal application of lidocaine cream 5% for 20 minutes before probe insertion. After probe insertion and prior to biopsy, a periprostatic nerve block was performed with 10 mL of 1% Lidocaine (5 mL on each side).
  Interventions: Procedure: Trans rectal ultrasound guided prostate biopsy; Procedure: Trans rectal ultrasound; Procedure: Prostate biopsy; Procedure: Periprostatic nerve block
- External Anal plus intrarectal - 5 minutes exposure (Active Comparator): Anal application plus intrarectal application of 5% lidocaine cream for 5 minutes before probe insertion.
  After probe insertion and prior to biopsy, a periprostatic nerve block was performed with 10 mL of 1% Lidocaine (5 mL on each side).
  Interventions: Procedure: Trans rectal ultrasound guided prostate biopsy; Procedure: Trans rectal ultrasound; Procedure: Prostate biopsy; Procedure: Periprostatic nerve block
- External Anal plus intrarectal - 10 minutes exposure (Active Comparator): Anal application plus intrarectal application of 5% lidocaine cream for 10 minutes before probe insertion.
  After probe insertion and prior to biopsy, a periprostatic nerve block was performed with 10 mL of 1% Lidocaine (5 mL on each side).
  Interventions: Procedure: Trans rectal ultrasound guided prostate biopsy; Procedure: Trans rectal ultrasound; Procedure: Prostate biopsy; Procedure: Periprostatic nerve block
- External Anal plus intrarectal - 20 minutes exposure (Active Comparator): Anal application plus intrarectal application of 5% lidocaine cream for 20 minutes before probe insertion.
  After probe insertion and prior to biopsy, a periprostatic nerve block was performed with 10 mL of 1% Lidocaine (5 mL on each side).
  Interventions: Procedure: Trans rectal ultrasound guided prostate biopsy; Procedure: Trans rectal ultrasound; Procedure: Prostate biopsy; Procedure: Periprostatic nerve block
- Control group (Sham Comparator): No anal application of lidocaine cream prior to probe insertion. After probe insertion and prior to biopsy, a periprostatic nerve block was performed with 10 mL of 1% Lidocaine (5 mL on each side).
  Interventions: Procedure: Trans rectal ultrasound guided prostate biopsy; Procedure: Trans rectal ultrasound; Procedure: Prostate biopsy; Procedure: Periprostatic nerve block

INTERVENTIONS:
Procedure: Trans rectal ultrasound guided prostate biopsy — The investigators checked visual analogue scale of pain at different time periods: prior to probe insertion, during probe insertion. during probe manipulation in the rectum, during performance of periprostatic nerve block, during actual biopsy collection and at termination of procedure.
Procedure: Trans rectal ultrasound — Performing a prostate biopsy using a transrectal ultrasound probe - the BK pro focus 2202 transrectal ultrasound and the 8808 bi-plane transrectal probe
  Other Names: BK pro focus 2202 transrectal ultrasound and the 8808 bi-plane transrectal probe
Procedure: Prostate biopsy — Prostate biopsy guided by a transrectal ultrasound with an 18 gauge needle
Procedure: Periprostatic nerve block — Performing a bilateral peri-prostatic nerve block with 10 mL of 1% lidocaine (5 mL on each side)

SUMMARY:
Transrectal ultrasound guided prostate biopsy is performed with a periprostatic nerve block to the neurovascular bundle bilaterally. This does not reduce the pain due to probe insertion and manipulation prior to nerve blockage.

Our study goal is to assess whether topical analgesia would reduce pain during the early stages of the procedure.

DETAILED DESCRIPTION:
Prospective, randomized controlled study. Patients signed an informed consent form. Exclusion criteria were Lidocaine allergy or pre-planned general anesthesia.

Patients were randomized into 6 groups: (1) nerve block with 5 ml 1% lidocaine for each neurovascular bundle + perianal topical application of 10 ml 5% lidocaine cream; (2) as in (1) plus application of 10 ml 5% lidocaine cream evenly on rectal walls. For each approach exposure times of 5, 10 and 20 minutes were allowed, all together 6 groups plus a control group of patients who received periprostatic nerve block only. A 0-10 Visual analogue scale (VAS) was filled by the patients at 5 time points: immediately after probe insertion, during probe manipulation and prostate assessment, immediately following neurovascular bundle nerve blockage, after prostate biopsies and a global pain estimation of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Males referred to TRUSGBx due to elevated prostate specific antigen (PSA)
* Abnormal findings on digital rectal examination (DRE)
* Repeat biopsies as part of Active Surveillance (AS)
* Continuously elevated PSA levels despite prior negative for malignancy biopsies
* Previous histological findings of significant HGPIN were enrolled

Exclusion Criteria:

* Known sensitivity to Lidocaine
* Pre-planned biopsy under general anesthesia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only those patients requiring a prostate biopsy
Enrollment: 284 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Pain level before probe insertion | Before transrectal ultrasound probe insertion
  Self reported by the patient using a 0-10 visual analogue scale. 0 being no pain at all, 10 being worst pain imaginable.
Pain level at TRUS probe insertion | During transrectal ultrasound probe insertion into the rectum (defined as beginning of procedure)
  Self reported by the patient using a 0-10 visual analogue scale. 0 being no pain at all, 10 being worst pain imaginable.
Pain level during TRUS probe manipulation in the rectum | During transrectal ultrasound probe manipulation in the rectum (estimated at 0-2 minutes length)
  Self reported by the patient using a 0-10 visual analogue scale. 0 being no pain at all, 10 being worst pain imaginable.
Pain level during periprostatic nerve block | During periprostatic nerve block (rectal wall puncture with needle, estimated at 2-3 minutes after beginning of procedure)
  Self reported by the patient using a 0-10 visual analogue scale. 0 being no pain at all, 10 being worst pain imaginable.
Pain level during biopsy collection | During biopsy collection using an 18-gauge needle (estimated at 3-10 minutes from beginning of procedure)
  Self reported by the patient using a 0-10 visual analogue scale. 0 being no pain at all, 10 being worst pain imaginable.
Pain level at termination of procedure | At termination of procedure (total estimated length of procedure is 10 minutes).
  Self reported by the patient using a 0-10 visual analogue scale. 0 being no pain at all, 10 being worst pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Ben Zvi, Study Chair — Assaf Harofeh Medical Center ethical committee for experiments in humans

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lee C, Woo HH. Current methods of analgesia for transrectal ultrasonography (TRUS)-guided prostate biopsy -- a systematic review. BJU Int. 2014 Mar;113 Suppl 2:48-56. doi: 10.1111/bju.12433. PMID 24053451
- [Result] Tiong HY, Liew LC, Samuel M, Consigliere D, Esuvaranathan K. A meta-analysis of local anesthesia for transrectal ultrasound-guided biopsy of the prostate. Prostate Cancer Prostatic Dis. 2007;10(2):127-36. doi: 10.1038/sj.pcan.4500935. Epub 2007 Jan 9. PMID 17211441
- [Result] Wang J, Wang L, Du Y, He D, Chen X, Li L, Nan X, Fan J. Addition of intrarectal local analgesia to periprostatic nerve block improves pain control for transrectal ultrasonography-guided prostate biopsy: a systematic review and meta-analysis. Int J Urol. 2015 Jan;22(1):62-8. doi: 10.1111/iju.12595. Epub 2014 Aug 21. PMID 25141759
- [Result] Raber M, Scattoni V, Roscigno M, Deho F, Briganti A, Salonia A, Gallina A, Di Girolamo V, Montorsi F, Rigatti P. Topical prilocaine-lidocaine cream combined with peripheral nerve block improves pain control in prostatic biopsy: results from a prospective randomized trial. Eur Urol. 2008 May;53(5):967-73. doi: 10.1016/j.eururo.2007.09.005. Epub 2007 Sep 18. PMID 17904278
- [Result] Giannarini G, Autorino R, Valent F, Mogorovich A, Manassero F, De Maria M, Morelli G, Barbone F, Di Lorenzo G, Selli C. Combination of perianal-intrarectal lidocaine-prilocaine cream and periprostatic nerve block for pain control during transrectal ultrasound guided prostate biopsy: a randomized, controlled trial. J Urol. 2009 Feb;181(2):585-91; discussion 591-3. doi: 10.1016/j.juro.2008.10.002. Epub 2008 Dec 13. PMID 19084860
- [Result] Barcohana N, Duperon DF, Yashar M. The relationship of application time to EMLA efficacy. J Dent Child (Chic). 2003 Jan-Apr;70(1):51-4. PMID 12762609